CLINICAL TRIAL: NCT05056818
Title: Comparison of Synthetic Mammography Versus Full-Field Digital Mammography in Image Interpretation and Performance Metrics
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0974; NCI-2021-08879 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0974 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-09-01; First posted 2021-09-27 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical records): Patients' medical records and past imaging examinations are reviewed.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical records and past imaging examinations

SUMMARY:
This study compares synthetic mammography to full-field digital mammography in image interpretation and performance metrics. Digital breast tomosynthesis (DBT) has previously been found to be superior in performance to standard digital mammography in both screening and diagnostic settings for the early detection and improved diagnosis of breast cancers. DBT in combination with full-field digital mammography (FFDM) reduces recall rates and increases cancer detection rates relative to FFDM alone. Synthetic mammography is a 2-dimensional reconstructed image, using the dataset derived from the DBT acquisition, without requiring additional radiation dose. Collecting information from patients' medical records may help doctors analyze the characteristics, utility, and impact of synthetic mammography to compared to FFDM.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To analyze the characteristics, utility, and impact of synthetic mammography (SM), as compared with full-field digital mammography (FFDM).

OUTLINE:

Patients' medical records and past imaging examinations are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18 or older
* Consecutive cases in breast imaging center

Exclusion Criteria:

* Cases demonstrate administrative or technical errors (e.g. missing views, labeling inconsistent with report, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergo mammography between August 1, 2018 and August 31, 2020
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
To analyze the impact of synthetic mammography (SM), as compared with full-field digital mammography (FFDM | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ray C Mayo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org